CLINICAL TRIAL: NCT00681317
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD6280 When Given in Multiple Ascending Oral Doses in Healthy Male and Healthy Female Subjects of Non-child Bearing Potential
Brief Title: AZD6280 Multiple Ascending Dose Study
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, PhD, Medical Science Sr.Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D0850C00002
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteer
Keywords: Phase I; Pharmacokinetics
MeSH Terms: interventions — 4-amino-8-(2,5-dimethoxyphenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD6280

INTERVENTIONS:
Drug: AZD6280 — oral

SUMMARY:
This is a study to evaluate safety, tolerability, PK and PD effects of orally administered AZD6280 after single and repeated ascending doses.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be of non-child bearing potential.

Exclusion Criteria:

* Clinically significant illness within 2 weeks before the study start.
* Enrollment in another concurrent investigational study or intake of an investigational drug within 30 days or intake of an investigational drug within a period of 5 half lives of that drug prior to the screening visit
* Blood loss in excess of 200 mL within 30 days of Day -2, in excess of 400 mL within 90 days of Day -2, or in excess of 1200 mL within 1 year of Day -2
* Clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending oral doses of AZD7325 compared to placebo by assessment of adverse events, vital signs, physical examinations, laboratory parameters, and ECGs | Assessments are made at each visit, at least daily, during the study.

SECONDARY OUTCOMES:
Evaluation and characterization of the pharmacokinetics of AZD6280 | Blood samples will be taken during the study.
Evaluation of the pharmacodynamic effects of AZD6280 | Test batteries will be performed at specified times both before and following study drug administration
Identification of genes that influence the disposition, efficacy, safety and tolerability of AZD6280. | A single blood sample will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvan J. Hurewitz, MD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, US
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States